CLINICAL TRIAL: NCT01260584
Title: The Influence of Smoking Status on the Pharmacokinetics and Pharmacodynamics of Prasugrel and Clopidogrel in Aspirin-treated Subjects With Stable Coronary Artery Disease
Brief Title: The Influence of Smoking Status on Prasugrel and Clopidogrel Treated Subjects Taking Aspirin and Having Stable Coronary Artery Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CS747S-B-U4002
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Results first posted 2012-12-12 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2012-11

CONDITIONS: Coronary Artery Disease
Keywords: thienopyridine; antiplatelet; prasugrel; clopidogrel
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel (Experimental): Prasugrel 10 mg film-coated tablet daily dose × 10 days. To maintain blinding, placebo film-coated tablets matching clopidogrel in appearance will be given daily × 10 days to subjects in the prasugrel treatment group. In addition, aspirin 81 mg to 325 mg daily will be taken.
  Interventions: Drug: Prasugrel
- Clopidogrel (Active Comparator): Clopidogrel 75 mg film-coated tablet daily dose x 10 days To maintain blinding, placebo film-coated tablets matching prasugrel in appearance will be given daily × 10 days to subjects in the clopidogrel treatment group. In addition, aspirin 81 mg to 325 mg daily will be taken.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — One 10 mg film-coated, oral tablet daily x 10 days. In addition, aspirin 81 mg to 325 mg daily will be taken.
  Other Names: Effient
  Arms: Prasugrel
Drug: Clopidogrel — One 75 mg film-coated, oral tablet daily x 10 days. In addition, aspirin 81 mg to 325 mg daily will be taken.
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
This study is being conducted to determine if smoking will influence the platelet aggregation inhibition ability of clopidogrel and prasugrel. It will also determine if smoking has any effect on the plasma concentrations of the active metabolite of prasugrel and the active and inactive metabolites of clopidogrel.

The primary hypothesis is that smoking status will influence the antiplatelet effects and active metabolite concentrations of clopidogrel but will have no impact on prasugrel's antiplatelet effects or active metabolite concentrations.

DETAILED DESCRIPTION:
Subjects will be stratified according to smoking status prior to being randomized to 1 of the 2 treatment sequences: prasugrel 10 mg daily for 10 days followed by clopidogrel 75 mg daily for 10 days or clopidogrel 75 mg daily for 10 days followed by prasugrel 10 mg daily for 10 days. There will be a 14-day Washout Period between Active Treatment Period 1 (when subjects receive the first drug of the sequence) and the second Active Treatment Period 2 (Period 3) (when subjects receive the second drug of the sequence). All subjects will remain on the same dose of aspirin from baseline throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects > or = 18 years and <75 years of age;
* Weight > or = 60 kg;
* On aspirin therapy (81 mg to 325 mg daily) at the time of screening and able to maintain a consistent aspirin dosing regimen from the baseline visit through the final study visit;
* Subjects who do not have contraindications for a thienopyridine (ie, prasugrel, clopidogrel, or ticlopidine) and have a history of stable atherosclerosis represented by CAD, defined as any of the following:

  * Chronic stable angina;
  * Documented prior ACS event > or = 30 days before screening and not currently prescribed or currently on thienopyridine therapy;
  * Previous coronary revascularization including percutaneous transluminal coronary angioplasty, stent, or coronary artery bypass graft;
  * Coronary Artery Disease (> or = 40% obstruction) in at least one coronary vessel after angiography;
  * Documented history of positive stress test; or
  * High coronary artery calcium score (> or = 90th percentile for age and gender) determined by cardiac computed tomography scan;
* Current smokers who smoke > or = ½ pack per day of cigarettes with a NicAlert™ level of 6;
* Non-smokers with a NicAlert level of 0, 1, or 2;
* Female subjects who meet one of the following:

  * Women of childbearing potential with a negative serum pregnancy test at screening, who are not breastfeeding, do not plan to become pregnant during the study, and agree to use an approved method of birth control during the study. Approved methods of birth control are intrauterine device, diaphragm plus spermicide, or female condom plus spermicide. Abstinence, partner's use of condoms, partner's vasectomy, and hormonal contraceptives are NOT acceptable methods of contraception;
  * Women who have been postmenopausal for at least 1 year or have had a hysterectomy, bilateral salpingo-oophorectomy, or tubal ligation at least 6 months prior to signing the Informed Consent Form (ICF); and
* Subjects with a competent mental condition to provide written informed consent before entering the study.

Exclusion Criteria:

* Subjects who received a bare metal stent and/or a drug-eluting stent within the last 12 months;
* Subjects who have had an angiogram < or = 7 days before randomization;
* Any other formal indication for the use of a thienopyridine;
* Subjects with a history of refractory ventricular arrhythmias;
* Subjects with a history of an implantable defibrillator device;
* Subjects with a history or evidence of congestive heart failure (New York Heart Association Class III or above) within 6 months prior to screening;
* Subjects with significant hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg) at either the time of screening or baseline assessment;
* Bleeding risk exclusion criteria:

  * Any known contraindication to treatment with an anticoagulant or antiplatelet agent;
  * Prior history or clinical suspicion of cerebral vascular malformations, intracranial tumor, transient ischemic attack, or stroke, or recent history (within 3 months) of head trauma;
  * Prior history or presence of significant bleeding disorders (eg, hematemesis, melena, severe or recurrent epistaxis, hemoptysis, hematuria, or intraocular bleeding);
  * History (within the last 5 years) or presence of gastric ulcers. Previous history of duodenal ulcer is acceptable but must have been successfully surgically or medically treated with no further evidence of disease in the past 6 months (from screening);
  * Prior history of abnormal bleeding tendency (ie, prolonged bleeding on dental extraction, tonsillectomy, or previous surgical procedure);
  * Known prior history or presence of thrombocytopenia (platelet count <100,000/mm3) or thrombocytosis (platelet count >500,000/mm3) or recent history (within 6 months) of hemoglobin <10 mg/dL;
  * International normalized ratio (INR) >1.5 or activated partial thromboplastin time (aPTT) > upper limit of normal (ULN) of laboratory reference range at screening;
  * History of major surgery, severe trauma, fracture, or organ biopsy within 3 months prior to enrollment;
* Prior/concomitant therapy exclusion criteria:

  * Subjects taking prasugrel, clopidogrel, ticlopidine, cilostazol, dipyridamole, warfarin, heparin, direct thrombin inhibitors, or GPIIb/IIIa inhibitors < or = 10 days prior to randomization or during study participation;
  * Use (or planned use) of fibrinolytic agents within 30 days before screening or during study participation;
  * Subjects receiving treatment with nonsteroidal anti-inflammatory drugs or cyclooxygenase-2 inhibitors exceeding 3 doses per week;
  * Subjects taking proton pump inhibitors (eg, lansoprazole, esomeprazole, omeprazole, pantoprazole, or rabeprazole) < or = 10 days prior to randomization or during study participation;
  * Use or planned use of any herbal supplements < or = 10 days prior to randomization or during study participation;
  * Use or planned use of the following strong inhibitors of various CYP pathways < or =10 days prior to randomization or during study participation: ciprofloxacin, cimetidine, fluvoxamine, estradiol, ethinylestradiol, fluconazole, amiodarone, indinavir, nelfinavir, ritonavir, saquinavir, clarithromycin, erythromycin, telithromycin, itraconazole, ketoconazole, fluconazole, nefazodone, or grapefruit-containing products;
  * Use or planned use of the following strong inducers of various CYP pathways < or = 10 days prior to randomization or during study participation: rifampin, barbiturates, carbamazepine, dexamethasone, or St. John's Wort;
  * Female subjects taking hormonal contraception or hormonal replacement therapy during study participation;
* General exclusion criteria:

  * Investigative site personnel directly affiliated with the study or immediate family of investigative site personnel directly affiliated with the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted;
  * Daiichi Sankyo or Eli Lilly employees;
  * Currently enrolled in, or discontinued within the last 30 days from, any clinical study involving an investigational drug or device;
  * Have previously completed or withdrawn from this study;
  * Women who are known to be pregnant and/or who receive a positive serum pregnancy test result, and/or who have given birth within the past 90 days, and/or who are breastfeeding;
  * Results of clinical laboratory tests at the time of screening that are judged to be clinically significant for the subject, as determined by the Investigator;
  * Known allergies or intolerance to aspirin and/or thienopyridines (prasugrel, clopidogrel, or ticlopidine);
  * Evidence of significant active neuropsychiatric disease, alcohol abuse, or drug abuse, in the Investigator's opinion;
  * Evidence of active hepatic disease or any of the following: positive human immunodeficiency virus antibodies; positive hepatitis C antibody; positive hepatitis B surface antigen; serum alanine transaminase, aspartate transaminase, or gamma-glutamyltransferase > or = 3 × ULN of laboratory reference range; or bilirubin > or = 2 × ULN of laboratory reference range at screening;
  * Subjects who are unwilling to make themselves available for the duration of the study and who will not abide by the research unit policy and procedure and study restrictions.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Gurbel, MD, Principal Investigator — Sinai Center for Thrombosis Research
Locations (3):
- United States (3):
  - Sanai Center for Thrombosis Research, Baltimore, Maryland
  - Medpace Clinical Pharmacology Unit, Cincinnati, Ohio
  - The Carl and Edyth Lindner Center for Research and Education at the Christ Hospital, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Gurbel PA, Bliden KP, Logan DK, Kereiakes DJ, Lasseter KC, White A, Angiolillo DJ, Nolin TD, Maa JF, Bailey WL, Jakubowski JA, Ojeh CK, Jeong YH, Tantry US, Baker BA. The influence of smoking status on the pharmacokinetics and pharmacodynamics of clopidogrel and prasugrel: the PARADOX study. J Am Coll Cardiol. 2013 Aug 6;62(6):505-12. doi: 10.1016/j.jacc.2013.03.037. Epub 2013 Apr 16. PMID 23602770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 4, double-blind, double-dummy, randomized, crossover study of male and female subjects with stable CAD, who are currently receiving aspirin and do not have contraindications for a thienopyridine.
Pre-assignment Details: Subjects will be stratified according to smoking status prior to being randomized to 1 of the 2 treatment sequences: prasugrel followed by clopidogrel or clopidogrel followed by prasugrel. There will be a 14-day Washout Period between Active Treatment Periods 1 and 2. All subjects will remain on the same dose of aspirin throughout the study.
Groups:
- Clopidogrel Then Prasugrel Smokers; Clopidogrel Then Prasugrel Non-Smokers: Clopidogrel 75 mg film-coated tablet daily dose x 10 days To maintain blinding, placebo film-coated tablets matching prasugrel in appearance will be given daily × 10 days to subjects in the clopidogrel treatment group. In addition, aspirin 81 mg to 325 mg daily will be taken.
  Prasugrel : One 10 mg film-coated, oral tablet daily x 10 days. In addition, aspirin 81 mg to 325 mg daily will be taken.
- Prasugrel Then Clopidogrel Smokers; Prasugrel Then Clopidogrel Non-Smokers: Prasugrel 10 mg film-coated tablet daily dose × 10 days. To maintain blinding, placebo film-coated tablets matching clopidogrel in appearance will be given daily × 10 days to subjects in the prasugrel treatment group. In addition, aspirin 81 mg to 325 mg daily will be taken.
  Clopidogrel : One 75 mg film-coated, oral tablet daily x 10 days. In addition, aspirin 81 mg to 325 mg daily will be taken.
Period: Period 1
Arm/Group | Clopidogrel Then Prasugrel Smokers | Clopidogrel Then Prasugrel Non-Smokers | Prasugrel Then Clopidogrel Smokers | Prasugrel Then Clopidogrel Non-Smokers
Started | 27 | 28 | 27 | 28
Completed | 27 | 28 | 25 | 27
Not Completed | 0 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Clopidogrel Then Prasugrel Smokers | Clopidogrel Then Prasugrel Non-Smokers | Prasugrel Then Clopidogrel Smokers | Prasugrel Then Clopidogrel Non-Smokers
Started | 27 | 28 | 25 | 27
Completed | 26 | 25 | 20 | 26
Not Completed | 1 | 3 | 5 | 1
Not completed — Protocol Violation | 0 | 2 | 3 | 1
Not completed — Adverse Event | 1 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clopidogrel Then Prasugrel Smokers | Clopidogrel Then Prasugrel Non-Smokers | Prasugrel Then Clopidogrel Smokers | Prasugrel Then Clopidogrel Non-Smokers | Total
Number analyzed (Participants) | 27 | 28 | 27 | 28 | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 20 | 24 | 17 | 79
  >=65 years | 9 | 8 | 3 | 11 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (8.19) | 59.6 (8.60) | 56.7 (8.03) | 61.9 (7.86) | 59.4 (8.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 9 | 7 | 31
  Male | 19 | 21 | 18 | 21 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 3 | 3 | 16
  Not Hispanic or Latino | 21 | 24 | 24 | 25 | 94
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 4 | 6 | 23
  White | 19 | 22 | 22 | 22 | 85
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 28 | 27 | 28 | 110
Weight [Mean (Standard Deviation); unit: kg] | 87.04 (15.243) | 92.45 (18.433) | 91.74 (20.109) | 99.91 (23.096) | 92.85 (19.740)
Height [Mean (Standard Deviation); unit: cm] | 172.3 (8.15) | 172.5 (10.95) | 172.5 (10.72) | 173.7 (8.17) | 172.8 (9.48)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.20 (3.945) | 31.12 (5.821) | 30.70 (5.131) | 32.94 (6.592) | 31.01 (5.562)
Body Mass Index Group [Number; unit: participants] — number participants less than 30 kilograms per square meter and number of participants greater than or equal to 30 kilograms per square meter
  participants
    <30 kg/m^2 | 19 | 10 | 13 | 10 | 52
    >=30 kg/m^2 | 8 | 18 | 14 | 18 | 58
Smoking History [Number; unit: participants]
  Never Smoked | 0 | 14 | 0 | 11 | 25
  Currently Smoke | 27 | 0 | 27 | 0 | 54
  Formerly Smoked | 0 | 14 | 0 | 17 | 31
Alcohol Usage [Number; unit: participants]
  Never consumed | 6 | 9 | 8 | 8 | 31
  Currently consumes | 17 | 16 | 13 | 15 | 61
  Formerly consumed | 4 | 3 | 6 | 5 | 18
Cardiovascular history [Number; unit: participants] — Individual categories should not add up to equal total number participants in each arm.
  participants
    Diabetes mellitus | 5 | 9 | 8 | 9 | 31
    Hypertension | 19 | 16 | 21 | 20 | 76
    Hyperlipidemia | 26 | 24 | 26 | 27 | 103
    Peripheral artery disease | 3 | 0 | 5 | 2 | 10
CYP2C19 Phenotype Metabolic Rate [Number; unit: participants]
  Poor | 0 | 0 | 0 | 2 | 2
  Intermediate | 5 | 4 | 6 | 4 | 19
  Extensive | 18 | 23 | 20 | 22 | 83
  Ultrarapid | 3 | 1 | 1 | 0 | 5
  not reported | 1 | 0 | 0 | 0 | 1
CYP2C19 Phenotype Metabolic Extent [Number; unit: participants]
  Extensive metabolizers | 21 | 24 | 21 | 22 | 88
  Reduced metabolizers | 5 | 4 | 6 | 6 | 21
  Missing | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Inhibition of Platelet Aggregation (IPA) in Prasugrel-treated and Clopidogrel-treated Smokers and Non-smokers Following 9 Days of Maintenance Therapy.
Description: IPA will be measured by the Accumetrics P2Y12 Assay Device. Response will be assessed in P2Y12 Reaction Units and as Platelet Reactivity Index (vasodilator-stimulated phosphoprotein assay).
Time Frame: Baseline to day 10 for Active Treatment Periods 1 and 2
Population: 1 prasugrel smoker was unevaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: percentage of device derived inhibition
Groups:
- Prasugrel Smokers: participants who currently smoke while receiving prasugrel as test medication during study
- Prasugrel Non-Smokers: participants who do not currently smoke while receiving prasugrel as test medication during study
- Clopidogrel Smokers: participants who currently smoke while receiving clopidogrel as test medication during study
- Clopidogrel Non-Smokers: participants who do not currently smoke while receiving clopidogrel as test medication during study
Arm/Group | Prasugrel Smokers | Prasugrel Non-Smokers | Clopidogrel Smokers | Clopidogrel Non-Smokers
Number analyzed (Participants) | 50 | 52 | 47 | 54
percentage of device derived inhibition | 70.3 (2.91) | 65.6 (2.86) | 38.6 (3.01) | 30.9 (2.81)
Statistical Analysis 1: Comparison: Clopidogrel Smokers vs Clopidogrel Non-Smokers; For the sample size calculations for the co-primary endpoints, no Type 1 error rate was adjusted and both co-primary endpoints will be tested at the 0.05 level; Test type: Superiority or Other; p = 0.0624, Mixed Models Analysis; Mean Difference (Final Values) = 7.7, 95% CI 2-sided [-0.4 to 15.8], Standard Error of Mean 4.11
Statistical Analysis 2: Comparison: Prasugrel Smokers vs Clopidogrel Smokers; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 31.8, 95% CI 2-sided [25.1 to 38.4], Standard Error of Mean 3.35
Statistical Analysis 3: Comparison: Prasugrel Smokers vs Prasugrel Non-Smokers; Test type: Superiority or Other; p = 0.2440, Mixed Models Analysis; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [-3.3 to 12.8], Standard Error of Mean 4.08
Statistical Analysis 4: Comparison: Prasugrel Non-Smokers vs Clopidogrel Non-Smokers; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 34.7, 95% CI 2-sided [28.4 to 41.0], Standard Error of Mean 3.17
Statistical Analysis 5: Comparison: Prasugrel Non-Smokers vs Clopidogrel Smokers; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 27.0, 95% CI 2-sided [18.8 to 35.2], Standard Error of Mean 4.14

2. Secondary Outcome: Assessment of P2Y12 Reaction Units (PRU) by Treatment and Smoking Status
Description: Day 10 occurs in each treatment period at which time data collections are made. 12.1.4. Responders and Poor Responders
  Numerous studies have established an association between high on-treatment platelet reactivity with clopidogrel and an increased risk for post-PCI ischemic events. In this study, the percentages of "responders" and "poor responders" following treatment with prasugrel and clopidogrel were compared. Poor responders were defined based on an Accumetrics VerifyNow PRU >235 and a VASP PRI >50%, as assessed 24 hours after the 9th maintenance dose.
Time Frame: Day 10 for Active Treatment Periods 1 and 2
Population: 1 prasugrel smoker was unevaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: P2Y12 reaction unit
Arm/Group | Prasugrel Smokers | Prasugrel Non-Smokers | Clopidogrel Smokers | Clopidogrel Non-Smokers
Number analyzed (Participants) | 50 | 52 | 47 | 54
P2Y12 reaction unit | 85.1 (8.99) | 106.3 (8.73) | 178.9 (9.26) | 215.1 (8.59)
Statistical Analysis 1: Comparison: Clopidogrel Smokers vs Clopidogrel Non-Smokers; Test type: Superiority or Other; p = 0.0048, Mixed Models Analysis; Mean Difference (Final Values) = -36.2, 95% CI 2-sided [-61.1 to -11.2], Standard Error of Mean 12.65
Statistical Analysis 2: Comparison: Prasugrel Smokers vs Clopidogrel Smokers; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -93.8, 95% CI 2-sided [-116.7 to -71.0], Standard Error of Mean 11.54
Statistical Analysis 3: Comparison: Prasugrel Smokers vs Prasugrel Non-Smokers; Test type: Superiority or Other; p = 0.0924, Mixed Models Analysis; Mean Difference (Final Values) = -21.2, 95% CI 2-sided [-45.9 to 3.5], Standard Error of Mean 12.53
Statistical Analysis 4: Comparison: Prasugrel Non-Smokers vs Clopidogrel Non-Smokers; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -108.8, 95% CI 2-sided [-130.3 to -87.3], Standard Error of Mean 10.85
Statistical Analysis 5: Comparison: Prasugrel Non-Smokers vs Clopidogrel Smokers; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -72.6, 95% CI 2-sided [-97.8 to -47.5], Standard Error of Mean 12.73

3. Secondary Outcome: Assessment of Vasodilator Stimulated Phosphoprotein (VASP) by Treatment and Smoking Status
Description: Day 10 occurs in each treatment period at which time data collections are made. Numerous studies have established an association between high on-treatment platelet reactivity with clopidogrel and an increased risk for post-PCI ischemic events. In this study, the percentages of "responders" and "poor responders" following treatment with prasugrel and clopidogrel were compared. Poor responders were defined based on an Accumetrics VerifyNow PRU >235 and a VASP PRI >50%, as assessed 24 hours after the 9th maintenance dose.
Time Frame: Day 10 for Active Treatment Periods 1 and 2
Population: 1 prasugrel smoker was unevaluable for this measure.
Measure: Least Squares Mean (Standard Error); unit: % vasodilator stimulated phosphoprotein
Arm/Group | Prasugrel Smokers | Prasugrel Non-Smokers | Clopidogrel Smokers | Clopidogrel Non-Smokers
Number analyzed (Participants) | 50 | 52 | 47 | 54
% vasodilator stimulated phosphoprotein | 25.4 (2.64) | 31.2 (2.59) | 48.1 (2.73) | 55.7 (2.54)
Statistical Analysis 1: Comparison: Clopidogrel Smokers vs Clopidogrel Non-Smokers; Test type: Superiority or Other; p = 0.0423, Mixed Models Analysis; Mean Difference (Final Values) = -7.6, 95% CI 2-sided [-15.0 to -0.3], Standard Error of Mean 3.72
Statistical Analysis 2: Comparison: Prasugrel Smokers vs Clopidogrel Smokers; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -22.7, 95% CI 2-sided [-29.0 to -16.4], Standard Error of Mean 3.19
Statistical Analysis 3: Comparison: Prasugrel Smokers vs Prasugrel Non-Smokers; Test type: Superiority or Other; p = 0.1184, Mixed Models Analysis; Mean Difference (Final Values) = -5.8, 95% CI 2-sided [-13.1 to 1.5], Standard Error of Mean 3.70
Statistical Analysis 4: Comparison: Prasugrel Non-Smokers vs Clopidogrel Non-Smokers; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -24.5, 95% CI 2-sided [-30.5 to -18.5], Standard Error of Mean 3.02
Statistical Analysis 5: Comparison: Prasugrel Non-Smokers vs Clopidogrel Smokers; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = -16.9, 95% CI 2-sided [-24.3 to -9.5], Standard Error of Mean 3.76

4. Secondary Outcome: Responder Rate by Treatment and Smoking Status Based on P2Y12 Reaction Units (PRU) <= 235
Time Frame: Day 10 for Active Treatment Periods 1 and 2
Population: 1 prasugrel smoker participant was not evaluable for this measure.
Measure: Number; unit: % participants with PRU <=235
Arm/Group | Prasugrel Smokers | Prasugrel Non-Smokers | Clopidogrel Smokers | Clopidogrel Non-Smokers
Number analyzed (Participants) | 50 | 52 | 47 | 54
% participants with PRU <=235 | 98.0 | 96.2 | 76.6 | 61.1
Statistical Analysis 1: Comparison: Clopidogrel Smokers vs Clopidogrel Non-Smokers; Test type: Superiority or Other; p = 0.1331, Regression, Logistic; Odds Ratio (OR) = 2.06, 95% CI 2-sided [0.80 to 5.32]
Statistical Analysis 2: Comparison: Prasugrel Smokers vs Prasugrel Non-Smokers; Test type: Superiority or Other; p = 0.5813, Regression, Logistic; Odds Ratio (OR) = 1.99, 95% CI 2-sided [0.17 to 23.65]
Statistical Analysis 3: Comparison: Prasugrel Smokers vs Clopidogrel Smokers; Test type: Superiority or Other; p = 0.0127, Regression, Logistic; Odds Ratio (OR) = 16.54, 95% CI 2-sided [1.85 to 148.23]
Statistical Analysis 4: Comparison: Prasugrel Non-Smokers vs Clopidogrel Non-Smokers; Test type: Superiority or Other; p = 0.0013, Regression, Logistic; Odds Ratio (OR) = 17.11, 95% CI 2-sided [3.13 to 93.65]

5. Secondary Outcome: Responder Rate by Treatment and Smoking Status Based on Platelet Reactivity Index (PRI) <= 50%
Description: Numerous studies have established an association between high on-treatment platelet reactivity with clopidogrel and an increased risk for post-PCI ischemic events. In this study, the percentages of "responders" and "poor responders" following treatment with prasugrel and clopidogrel were compared. Poor responders were defined based on an Accumetrics VerifyNow PRU >235 and a VASP PRI >50%, as assessed 24 hours after the 9th maintenance dose.
Time Frame: Day 10 for Active Treatment Periods 1 and 2
Population: 1 prasugrel smoker participant was not evaluable for this measure.
Measure: Number; unit: % participants with PRI <=50%
Arm/Group | Prasugrel Smokers | Prasugrel Non-Smokers | Clopidogrel Smokers | Clopidogrel Non-Smokers
Number analyzed (Participants) | 50 | 52 | 47 | 54
% participants with PRI <=50% | 96.0 | 82.7 | 51.1 | 44.4
Statistical Analysis 1: Comparison: Clopidogrel Smokers vs Clopidogrel Non-Smokers; Test type: Superiority or Other; p = 0.5684, Regression, Logistic; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.49 to 3.67]
Statistical Analysis 2: Comparison: Prasugrel Smokers vs Prasugrel Non-Smokers; Test type: Superiority or Other; p = 0.0447, Regression, Logistic; Odds Ratio (OR) = 6.70, 95% CI 2-sided [1.05 to 42.92]
Statistical Analysis 3: Comparison: Prasugrel Smokers vs Clopidogrel Smokers; Test type: Superiority or Other; p = 0.0003, Regression, Logistic; Odds Ratio (OR) = 58.64, 95% CI 2-sided [6.80 to 505.58]
Statistical Analysis 4: Comparison: Prasugrel Non-Smokers vs Clopidogrel Non-Smokers; Test type: Superiority or Other; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 11.71, 95% CI 2-sided [2.95 to 46.52]

6. Secondary Outcome: Characterization of the Pharmacokinetics (PK) Area Under Curve (AUC)(0-Last) of the Active Metabolite of Prasugrel and the Active Metabolite of Clopidogrel in Smokers and Non-smokers
Description: Blood samples for determination of plasma concentrations of the prasugrel active metabolite, clopidogrel active metabolite, and clopidogrel inactive metabolite will be collected following the administration of the 10th (last) maintenance dose of each of the 2 Active Treatment Periods at 0.5, 1, 2, 4, and 6 hours post-dose.
Time Frame: After dose on Day 10 of Active Treatment Periods 1 and 2
Population: 1 Clopidogrel smoker participant was not evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Prasugrel Smokers | Prasugrel Non-Smokers | Clopidogrel Smokers | Clopidogrel Non-Smokers
Number analyzed (Participants) | 51 | 52 | 46 | 54
hr*ng/mL | 53.7 (41.2) | 48.1 (52.0) | 19.9 (55.8) | 16.2 (87.4)
Statistical Analysis 1: Comparison: Prasugrel Smokers vs Prasugrel Non-Smokers; Prasugrel active metabolite R-138727; Test type: Superiority or Other; Mixed Models Analysis; Risk Ratio (RR) = 110.7, 90% CI 2-sided [93.7 to 130.8]
Statistical Analysis 2: Comparison: Clopidogrel Smokers vs Clopidogrel Non-Smokers; active metabolite R-130964; Test type: Superiority or Other; Mixed Models Analysis; Risk Ratio (RR) = 118.4, 90% CI 2-sided [99.8 to 140.4]

7. Secondary Outcome: Characterization of the Pharmacokinetics (PK) Cmax of the Active Metabolite of Prasugrel and the Active Metabolite of Clopidogrel in Smokers and Non-smokers
Time Frame: After dose on Day 10 of Active Treatment Periods 1 and 2
Population: 1 clopidogrel smoker was not evaluable for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Prasugrel Smokers | Prasugrel Non-Smokers | Clopidogrel Smokers | Clopidogrel Non-Smokers
Number analyzed (Participants) | 51 | 52 | 46 | 54
ng/mL | 42.9 (66.1) | 35.9 (80.7) | 14.1 (84.3) | 10.8 (116.3)
Statistical Analysis 1: Comparison: Prasugrel Smokers vs Prasugrel Non-Smokers; Prasugrel active metabolite R-138727; Test type: Superiority or Other; Mixed Models Analysis; Risk Ratio (RR) = 117.9, 90% CI 2-sided [94.4 to 147.3] — Estimation was based on the ratio of Geom. means between groups. Non-smoker is the denominator
Statistical Analysis 2: Comparison: Clopidogrel Smokers vs Clopidogrel Non-Smokers; Clopidogrel active metabolite R-130964; Test type: Superiority or Other; Mixed Models Analysis; Risk Ratio (RR) = 123.8, 90% CI 2-sided [98.6 to 155.4] — Estimation was based on the ratio of Geom. means between groups. Non-smoker is the denominator

ADVERSE EVENTS:
Description: 1 prasugrel non-smoker, 2 clopidogrel smokers, 1 clopidogrel non-smoker did not receive treatment in one period and were not determined to be "at-risk".
Groups:
- Prasugrel Non-Smokers: participants who do not currently smoke while receiving prasugrel as test medication during study. 1 participant who started the arm was not "at risk".
- Clopidogrel Smokers: participants who currently smoke while receiving clopidogrel as test medication during study. 2 participants who started this arm were not "At risk".
- Clopidogrel Non-Smokers: participants who do not currently smoke while receiving clopidogrel as test medication during study. 1 participant who started this arm was not "at risk".
Arm/Group | Prasugrel Smokers | Prasugrel Non-Smokers | Clopidogrel Smokers | Clopidogrel Non-Smokers
Serious Adverse Events (participants affected / at risk) | 4/54 | 0/55 | 0/50 | 0/54
Other Adverse Events (participants affected / at risk) | 5/54 | 6/55 | 10/50 | 6/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel Smokers (N=54) | Prasugrel Non-Smokers (N=55) | Clopidogrel Smokers (N=50) | Clopidogrel Non-Smokers (N=54)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel Smokers (N=54) | Prasugrel Non-Smokers (N=55) | Clopidogrel Smokers (N=50) | Clopidogrel Non-Smokers (N=54)
Vessel puncture site hemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal Dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reflects the following restrictive language in the Clinical Study Agreements: "If Daiichi Sankyo Inc. (DSI) identifies any of its confidential information as defined herein, it shall be deleted … Nothing in this publication section shall be taken as giving DSI any right of editorial control over any publication prepared by the Study Site."